CLINICAL TRIAL: NCT06554054
Title: A Randomized, Open Phase I Trial to Evaluate the Bioavailability, Pharmacokinetics, Pharmacodynamics, Safety and Tolerance of GZR18 Tablet and Evaluate the Effect of Meal Time on the Pharmacokinetics, Pharmacodynamics, Safety and Tolerance of GZR18 Tablet in Chinese Healthy Adult Subjects
Brief Title: A Study of GZR18 Tablet in Chinese Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GLP-CH1010
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Part A (single dose) (Experimental): Drug: GZR18 tablet Three single-dose cohorts of GZR18 tablet administered according to an ascending dose design. Progression to next dose will be based on safety evaluation. Sequential cohorts.
  Active Comparator: GZR18 injection Single-dose administered s.c. (under the skin).
  Interventions: Drug: GZR18
- Experimental: Part B (multiple dose) (Experimental): Drug:GZR18 tablet GZR18 tablet administered as two multiple dose cohorts, to test the different meal time effect.
  Parallel assignment
  Interventions: Drug: GZR18

INTERVENTIONS:
Drug: GZR18 — Oral administered the GZR18 tablet

SUMMARY:
The aim of the trial is to investigate the the bioavailability, pharmacokinetics, pharmacodynamics, safety and tolerance of single and multiple doses of GZR18 tablet in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects sign informed consent voluntarily.
2. Age 18-55 at screening (both included)，male or female（male only for part A）.
3. At screening, 20.0 kg/m2 ≤ BMI ≤ 24.9 kg/m2, body weight≥54.0 kg.
4. Female subjects were HCG negative at screening and baseline

Exclusion Criteria:

1. Female subjects who are pregnant or lactating at screening.
2. History of drug abuse within 1 year prior to screening, with a positive drug abuse screening result at screening or before dosing.
3. Abnormal fasting blood glucose at screening, or impaired glucose tolerance, or history of hypoglycemia within 3 months prior to screening.
4. History of the following diseases with a definite diagnosis within 6 months prior to screening: cardiovascular disease, hematologic disease, respiratory disease, abnormal liver function due to acute and chronic hepatitis or other reasons, abnormal renal function, endocrine and metabolic system disease, neuropsychiatric disease, skin and subcutaneous tissue disease, musculoskeletal system disease, immune system disease, or the presence of other diseases that may interfere with the interpretation of study results.
5. Those who have any food allergies or special dietary requirements and cannot follow a uniform diet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-09 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
AE and SAE | 22 days and 35 days
  Incidence of Adverse Events and Severe Adverse Events
Relative bioavailability of GZR18 tablet | 22 days and 35 days
  Fr =AUC0-t(GZR18 tablets)/AUC0-t(GZR18 injection)×100%
ADA and NAb | 22 days and 35 days
  Anti-Drug Antibody (ADA) and Neutralizing Antibody (Nab)

SECONDARY OUTCOMES:
Cmax | 22 days and 35 days
  Maximum plasma drug concentration
AUC0-t | 22 days and 35 days
  Area under the curve from 0 through the time of the last accurately measurable concentration
AUC0-24h | 22 days and 35 days
  Area under the curve from 0 h to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Min, Ph.D, Study Director — Gan & Lee Pharmaceuticals Co., Ltd
Locations (1):
- Study Site 01, Beijing, China